CLINICAL TRIAL: NCT03159715
Title: Internet-based Depression Treatment. Differential Efficacy of Different Specific Therapeutic Components: Behavioral Activation and Positive Psychology.
Brief Title: Internet-based Depression Treatment: Differential Efficacy of Different Therapeutic Components
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Jaume I (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2017-05-17; First posted 2017-05-19 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Depression
Keywords: Internet, Behavioral Activation, Positive Psychology
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-based Global Protocol (Experimental): Intervention group that carries out the Internet-based Global Protocol and receives therapist support.
  Interventions: Behavioral: Internet-based Global Protocol
- Internet-based Behavioral Activation Protocol (Experimental): Intervention group that carries out the Internet-based Behavioral Activation Protocol and receives therapist support.
  Interventions: Behavioral: Internet-based Behavioral Activation Protocol
- IInternet-based Positive Psychology Protocol (Experimental): Intervention group that carries out the Internet-based Positive Psychology Protocol and receives therapist support.
  Interventions: Behavioral: Internet-based Positive Psychology Protocol

INTERVENTIONS:
Behavioral: Internet-based Global Protocol — Internet-based Global Protocol is an Internet-based treatment which includes therapeutic components of evidence-based treatments for depression: Motivation, Psychoeducation, Cognitive Therapy, and Relapse Prevention. Furthermore, it incorporates a Behavioural Activation component (BA). The whole protocol stresses the importance and benefits of being active and remaining involved in life, values and goals. The program also includes a component of Positive Psychology (PP). It allows the individual to learn and practice adaptive ways to cope with depressive and anxiety symptoms and confront daily problems. It is a multimedia (video, image, etc.) interactive program designed for optimal use on the computer, but it can also be used on a tablet.
  Arms: Internet-based Global Protocol
Behavioral: Internet-based Behavioral Activation Protocol — Internet-based Behavioral Activation Protocol is an Internet-based treatment based on Behavioral Activation. It stresses the importance and benefits of being active and remaining involved in life, values and goals . It is a multimedia (video, image, etc.) interactive program designed for optimal use on the computer, but it can also be used on a tablet.
  Arms: Internet-based Behavioral Activation Protocol
Behavioral: Internet-based Positive Psychology Protocol — Internet-based Positive Psychology Protocol is an Internet-based treatment based on Positive Psychology, offering strategies to promote and enhance positive mood. It is an Internet-based treatment based on Positive Psychology. It is a multimedia (video, image, etc.) interactive program designed for optimal use on the computer, but it can also be used on a tablet.
  Arms: IInternet-based Positive Psychology Protocol

SUMMARY:
The objective of the present project is to study the differential effectiveness of three brief self-applied via the Internet interventions for mild to moderate depression: a global protocol composed of several therapeutic components (psychoeducation, cognitive restructuring, behavioral activation, positive psychology, and relapse prevention), a protocol just based on behavioral activation (BA), and a protocol just based on positive psychology (PP). The purpose is to know the specific contribution of each therapeutic components in the treatment of depression.

DETAILED DESCRIPTION:
Depression is one of the most important health problems worldwide, which generates important costs, both from the economic point of view as from the social and personal one. If not properly treated, it may become chronic and therefore interferes significantly in all areas of operation. Hence, one of the most important challenges within this scope is the design of new ways to apply treatments in a way that maximizes its therapeutic efficiency. Information and Communication Technologies (ICTs) have proven their utility as they are very useful in order to provide help to all those in need. It is a field of study very novel which will become more important in the short term. Several internationally renowned research groups have launched self-applied treatment programs through the Internet in order to address this issue. Results obtained so far are consistent and promising, and show these treatments as effective. However, these treatments have different therapeutic components and it is important to identify the specific contribution of each of them. Therefore, the objective of the present project is to study the differential effectiveness of three brief self-applied via the Internet interventions for mild to moderate depression: a global protocol composed of several therapeutic components (psychoeducation, cognitive restructuring, behavioral activation, positive psychology, and relapse prevention), a protocol just based on behavioral activation (BA), and a protocol just based on positive psychology (PP). A minimum of 192 participants diagnosed with mild to moderate depression symptoms will be randomly assigned to one of the three experimental conditions: an Internet-based global protocol composed of several therapeutic components (n=64); a Internet-based protocol based on BA (n=64), and an Internet-based program based on PP (n=64). Our hypothesis is that it is possible to progress and improve in the treatment of depression through intervention strategies applied through the Internet.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old.
* Having mild to moderate depression symptoms.
* Providing written, informed consent.
* Being able to understand and read Spanish.
* Having daily access to the Internet in their natural environment.

Exclusion Criteria:

* Being diagnosed a severe mental disorder (people with the following mental disorders will be excluded from the study: schizophrenia, bipolar disorder and personality disorders from clusters A and B).
* Being diagnosed an alcohol and/or substance dependence disorder.
* The presence of high suicidal risk.
* A medical disease or condition which prevent the participant from carry out the psychological treatment.
* Receiving another psychological treatment while the study is still ongoing.
* The increase and/or changes in the medication of participants receiving pharmacological treatment during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Change in the Beck Depression Inventory II (BDI-II) (Beck, Steer, & Brown, 1996) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The BDI-II is one of the most widely used questionnaires to evaluate the severity of depression in pharmacological and psychotherapy trials. It consists of 21 items about the different symptoms characterizing the major depression disorder, summed to obtain the total score, which can be a maximum of 63 points. The instrument has good internal consistency (Cronbach's alpha of 0.76 to 0.95) and a test-retest reliability of around 0.8.

SECONDARY OUTCOMES:
The Positive and Negative Affect Schedule (PANAS) (Watson, Clark y Tellegen, 1988; Sandín et al., 1999) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  The PANAS consists of 20 items that evaluate two independent dimensions: positive affect (PA) and negative affect (NA). The range for each scale (10 items on each) is from 10 to 50. The Spanish version has demonstrated high internal consistency (α = 0.89 and 0.91 for PA and NA in women, respectively, and α = 0.87 and 0.89 for PA and NA in men, respectively) in college students.
Overall Anxiety Severity and Impairment Scale (OASIS) Overall Depression Severity and Impairment Scale (ODSIS) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  OASIS consists of 5 items that measure the frequency and severity of anxiety, as well as the level of avoidance, work/ school/home interference, and social interference associated to anxiety. A psychometric analysis of the OASIS scale found good internal consistency (Cronbach's alpha = 0.80), test-retest reliability (k = 5.82) and convergent validity for this scale.
Overall Depression Severity and Impairment Scale (ODSIS) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  ODSIS is a self-report measure which consists of 5 items, evaluating experiences related to depression. ODSIS measures the frequency and severity of depression, as well as the level of avoidance, work/school/home interference, and social interference associated to depression.
Multicultural Quality of Life Index (MQLI) at pre, post intervention and at 3 and 12 months follow-ups. | Up to 12 months
  It is a self-administered questionnaire that uses 10 items to assess global perception of quality of life in addition to physical and emotional well-being, self-care, occupational, and interpersonal functioning, community and services support, and personal and spiritual fulfilment. The homogeneity of the questionnaire proved to be good, yielding a Cronbach's alpha coefficient of 0.79 and has applicability, reliability, and validity.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Mira, Phd, Principal Investigator — Universitat Jaume I; Cristina Botella, Professor, Study Director — Universitat Jaume I
Locations (1):
- University Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mira A, Breton-Lopez J, Garcia-Palacios A, Quero S, Banos RM, Botella C. An Internet-based program for depressive symptoms using human and automated support: a randomized controlled trial. Neuropsychiatr Dis Treat. 2017 Mar 31;13:987-1006. doi: 10.2147/NDT.S130994. eCollection 2017. PMID 28408833
- [Background] Karyotaki E, Riper H, Twisk J, Hoogendoorn A, Kleiboer A, Mira A, Mackinnon A, Meyer B, Botella C, Littlewood E, Andersson G, Christensen H, Klein JP, Schroder J, Breton-Lopez J, Scheider J, Griffiths K, Farrer L, Huibers MJ, Phillips R, Gilbody S, Moritz S, Berger T, Pop V, Spek V, Cuijpers P. Efficacy of Self-guided Internet-Based Cognitive Behavioral Therapy in the Treatment of Depressive Symptoms: A Meta-analysis of Individual Participant Data. JAMA Psychiatry. 2017 Apr 1;74(4):351-359. doi: 10.1001/jamapsychiatry.2017.0044. PMID 28241179
- [Background] Botella C, Mira A, Moragrega I, Garcia-Palacios A, Breton-Lopez J, Castilla D, Riera Lopez Del Amo A, Soler C, Molinari G, Quero S, Guillen-Botella V, Miralles I, Nebot S, Serrano B, Majoe D, Alcaniz M, Banos RM. An Internet-based program for depression using activity and physiological sensors: efficacy, expectations, satisfaction, and ease of use. Neuropsychiatr Dis Treat. 2016 Feb 23;12:393-406. doi: 10.2147/NDT.S93315. eCollection 2016. PMID 27042067
- [Background] Karyotaki E, Kleiboer A, Smit F, Turner DT, Pastor AM, Andersson G, Berger T, Botella C, Breton JM, Carlbring P, Christensen H, de Graaf E, Griffiths K, Donker T, Farrer L, Huibers MJ, Lenndin J, Mackinnon A, Meyer B, Moritz S, Riper H, Spek V, Vernmark K, Cuijpers P. Predictors of treatment dropout in self-guided web-based interventions for depression: an 'individual patient data' meta-analysis. Psychol Med. 2015 Oct;45(13):2717-26. doi: 10.1017/S0033291715000665. Epub 2015 Apr 17. PMID 25881626
- [Derived] Mira A, Diaz-Garcia A, Castilla D, Campos D, Romero S, Breton-Lopez J, Garcia-Palacios A, Banos R, Botella C. Protocol for a randomized controlled dismantling study of an internet-based intervention for depressive symptoms: exploring the contribution of behavioral activation and positive psychotherapy strategies. BMC Psychiatry. 2019 May 3;19(1):133. doi: 10.1186/s12888-019-2099-2. PMID 31053067
- See also: Description Laboratory of Psychology and Technology of the University Jaume I — http://www.labpsitec.uji.es
- See also: Description Web site of the intervention programs — http://psicologiaytecnologia.com